CLINICAL TRIAL: NCT03449706
Title: Accurate Staging of Immuno-virological Dynamics During Acute HIV Infection
Acronym: ACS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ACS
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: HIV; Seroconversion, HIV
Keywords: Reservoir
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Colon biopsy
  * Lymph node biopsy
  * Cerebrospinal fluids
  * Whole blood
  * Leukapheresis apherate
  * Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Early combination anti-retroviral treatment — Patients are started on treatment to supress the HIV virus in the phase of acute seroconversion.

SUMMARY:
In this prospective longitudinal study we aim to assess how immunologic and viral aspects of the human immunodeficiency virus (HIV) viral reservoir, established during early HIV infection and responsible for viral rebound at treatment interruption, evolve in individuals who start combination anti-retroviral therapy (cART) during acute seroconversion.

Recently infected patients will be selected based on Fiebig staging for an in depth sampling protocol at different timepoints during a 2 year follow up period. Colonbiopsies, lymphnode resection, lumbar puncture, leucapheresis and repeated peripheral venous blood-draws will be performed. Immunological, virological and genome expression analysis will be performed on the gathered samples.

ELIGIBILITY:
Inclusion Criteria:

* Documented recent HIV-1 infection, early diagnosis: clinical symptoms of acute seroconversion and incomplete Western Blot OR negative screening test within the past 6 months and incomplete Western Blot OR risk contact within the 3 months and presumable primo-infection with or without clinical symptoms and incomplete Western Blot
* Able and willing to provide written informed consent
* Ability to attend the complete schedule of assessments and patient visits for patients participating in option A schedule (described below), or ability to attend a partial schedule of assessments and patient visits for patients participating in option B (described below).
* Ability and willingness to have blood and tissue samples collected and stored indefinitely and used for various research purposes.

Exclusion Criteria:

* Previous or current history of opportunistic infection (AIDS defining events as defined in category C of the CDC clinical classification), consisting of chronic HIV-1 infection.
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (=HBV antigen or viral load negative and positive HBV surface antibody).
* Evidence of active HCV infection: HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry.
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* Current history of cancer.
* Pregnancy or breastfeeding.
* Any conditions, including psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant.
* Previous participation in a trial evaluating an immune modulating agent
* Abnormal laboratory tests results at screening: confirmed Hemoglobin <11g/dl for women and <12 g:dl for men/ confirmed platelet count < 100000/l / confirmed neutrophil count <1000/μl/ confirmed AST and/or ALT > 3xULN
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll a minimum of 30 patients and a maximum of 70 participants (Fiebig stages I - VI) in the study to establish a cohort of early treated patients. We aim at including at least 15 people with an incomplete Western Blot (Fiebig I->IV) and as a control we will also include patients with complete Western Blot and history of a semi-recent infection (Fiebig V-VI).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of virological and immunological parameters of the HIV reservoir in recently infected HIV positive patients that started treatment during acute seroconversion. | 10 years
  Virological, immunological and gene expression analysis on blood and tissue from in depth sampling.

SECONDARY OUTCOMES:
Evolution of microbiome in recently infected HIV positive patients that started treatment during acute seroconversion. | 10 years
  Microbiome analysis on stoolsamples.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT03449706/Prot_000.pdf
  • Informed Consent Form (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT03449706/ICF_001.pdf